CLINICAL TRIAL: NCT05744674
Title: A Phase Ⅱ Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Single Injection Intercostal Nerve Block With HR18034 for Postoperative Pain Management
Brief Title: Phase Ⅱ Study of Intercostal Nerve Block With HR18034 for Postsurgical Pain Management
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HR18034-203
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Thoracoscopic Lobectomy
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: HR18034 compared with active comparator
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR18034 (Experimental)
  Interventions: Drug: HR18034
- Ropivacaine Hydrochloride Injection (Active Comparator)
  Interventions: Drug: Ropivacaine Hydrochloride Injection

INTERVENTIONS:
Drug: HR18034 — HR18034 228mg/342mg/456mg
  Arms: HR18034
Drug: Ropivacaine Hydrochloride Injection — Ropivacaine Hydrochloride Injection 60mg/90mg/120mg
  Arms: Ropivacaine Hydrochloride Injection

SUMMARY:
Phase Ⅱ, randomized, double-blind, comparator-controlled study to evaluate the efficacy, safety and pharmacokinetics of single injection intercostal nerve block with HR18034 for postoperative pain management compared with ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Scheduled to undergo thoracoscopic lobectomy under general anesthesia.
3. Male or female, aged 18 years and older inclusive
4. Body mass index (BMI) 18-30 kg/m2 inclusive
5. American Society of Anesthesiologists (ASA) Physical Status Classification Ⅰ~Ⅱ

Exclusion Criteria:

1. Subjects with a history of new myocardial infarction or unstable angina within 6 months prior to randomization;
2. Subjects with a history of ischemic stroke or transient ischemic attack (TIA)
3. Subjects with a history of mental system diseases and cognitive dysfunction
4. Combination of other pain conditions that may affect postoperative pain assessment
5. Combination with ventilation disorders caused by airway or spinal anatomical factors, bronchiectasis, and severe chest adhesions on the surgical side
6. Clinically significant abnormal clinical laboratory test value
7. Allergic to a drug ingredient or component
8. Use of any of medications, which affect drug metabolism or analgesia evaluation, within 5 half-lives or as specified prior to the study surgical procedure
9. History of alcohol abuse or prescription and/or illicit drug abuse
10. Subjects with special diets (including tobacco, grapefruit and caffeine)
11. Pregnant or nursing women
12. No birth control during the specified period of time
13. Participated in clinical trials of other drugs (received experimental drugs)
14. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
AUC0-72 of the NRS-A (or cough) pain intensity scores. | 0 to 72 hours
  AUC of NRS pain intensity scores at activity (NRS-A) through 72 hours after the beginning of study drug administration.

SECONDARY OUTCOMES:
AUC of the NRS-A (or cough) pain intensity scores. | 0-12, 12-24,12-48, 12-72 hours
  AUC of NRS pain intensity scores at activity (NRS-A) or cough for time periods 0-12, 12-24, 12-48, 12-72 hours.
AUC of the NRS-R pain intensity scores. | 0-12, 12-24,12-48, 12-72, 0-72 hours
  AUC of NRS pain intensity scores at rest (NRS-R) for time periods 0-12, 12-24,12-48, 12-72, 0-72 hours.
Proportion of subjects who used no rescue opioid analgesic. | 0-24, 24-48, 48-72, 0-72 hours
  Proportion of subjects who used no rescue opioid analgesic through 0-24, 24-48, 48-72 and 0-72 hours after the beginning of study drug administration.
Total rescue analgesic consumption. | 0-24, 24-48, 48-72, 0-72 hours
  Total rescue analgesic consumption through 0-24, 24-48, 48-72 and 0-72 hours after the beginning of study drug administration.
Time to the first postoperative use of rescue opioid analgesics. | 0-72 hours
  Time to the first postoperative use of rescue opioid analgesics 0-72 hours after the beginning of study drug administration.
Subjects' satisfaction rating | 72 hours
  Subjects' satisfaction rating with postsurgical pain control at 72 hours.
Investigators' satisfaction rating | 72 hours
  Investigators' satisfaction rating with postsurgical pain control at 72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided